CLINICAL TRIAL: NCT00427284
Title: Effect of Eplerenone on Endothelial Function in Patients With Stable Coronary Heart Disease
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: EK 1033
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2011-12-23 (Estimated); Status verified 2011-12

CONDITIONS: Coronary Artery Disease
Keywords: Eplerenone auf die Endothelfunktion bei Patienten mit stabiler koronarer Herzkrankheit
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
The aim of the present study is to investigate wether endothelial dysfunction associated with stable coronary artery disease is altered by selective aldosterone antagonism with Eplerenone as potential anti-inflammatory drug versus placebo.

Additionally we hypothesize that selective aldosterone antagonism reduces systemic inflammatory response such as C-reactive proteine, oxidative stress and pro-inflammatory cytokines.

ELIGIBILITY:
Inclusion criteria:

* Male patients (> 30 years of age) with history of coronary artery disease (documented by coronary angiogram, nuclear imaging, positive stress test)
* Stable cardiovascular medication for at least 4 months Evaluation of the patients will take place at the Department of Internal Medicine, Cardiology, University Hospital Zurich.

Exclusion criteria:

* Evidence for myocardial infarction, unstable angina, stroke within 3 months prior to study entry
* coronary intervention/re-vascularisation procedure within 3 months prior to study entry
* long acting nitrates
* uncontrolled arterial hypertension, defined as RR>160/90 mmHg
* congestive heart failure (> NYHA I)
* Ejection fraction <50%
* AV-Block>I˚
* creatinine clearance <50 mL/min
* insulin-dependent diabetes mellitus
* type 2 diabetes with microalbuminuria
* age < 30 years
* anemia (Hb<10 g/dl)
* malignancy chronic infection
* smoking
* serum potassium >5.5 meq/L
* drug abuse
* potassium supplements or potassium-sparing diuretics (amiloride, spironolactone, or triamterene)
* concomitant use of strong inhibitors of CYP450 3A4 (e.g., ketoconazole, itraconazole)
* known history of Cushing disease or Morbus Addisons or diseases of the thyroid gland

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary heart disease
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2004-07

CONTACTS AND LOCATIONS:
Overall Officials: Frank Ruschitzka, Prof MD, Principal Investigator — University Hospital Zurich, Division of Cardiology
Locations (1):
- University Hospital Zurich, Division of Cardiology, Zurich, Canton of Zurich, Switzerland